CLINICAL TRIAL: NCT06286644
Title: Effect of Iso-alpha Acids and Xanthohumol on the Human Immune System
Brief Title: Hop Compounds on the Immune System (VH)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ina Bergheim, Principal Investigator, University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UVienna23
Record Dates: First submitted 2024-01-17; First posted 2024-02-29 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Response
MeSH Terms: interventions — xanthohumol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Xanthohumol (Experimental): Participants receive a study drink supplemented with Xanthohumol (0mg = Placebo; 0,125 mg; 0,375 mg or 0,75 mg soluble Xanthohumol)
  Interventions: Dietary Supplement: Xanthohumol
- Iso-alpha-Acids (Experimental): Participants receive a study drink supplemented with Xanthohumol (0 mg = Placebo; 15 mg, 45 mg or 90 mg Iso-alpha-Acids)
  Interventions: Dietary Supplement: Iso-alpha-Acids
- Xanthohumol/Iso-alpha-Acids (Experimental): Participants receive a study drink supplemented with Xanthohumol + Iso-alpha-Acids (0 mg = Placebo; 0,125 mg + 15 mg, 0,375 mg + 45 mg or 0,75 mg + 90 mg soluble Xanthohumol + Iso-alpha-Acids)
  Interventions: Dietary Supplement: Xanthohumol + Iso-alpha-Acids

INTERVENTIONS:
Dietary Supplement: Xanthohumol — Participants receive a study drink supplemented with Xanthohumol (0 mg = Placebo, 0,125 mg, 0,375 mg or 0,75 mg soluble Xanthohumol)
  Arms: Xanthohumol
Dietary Supplement: Iso-alpha-Acids — Participants receive a study drink supplemented with Iso-alpha-Acids (0 mg = Placebo, 15 mg, 45 mg or 90 mg Iso-alpha-Acids)
  Arms: Iso-alpha-Acids
Dietary Supplement: Xanthohumol + Iso-alpha-Acids — Participants receive a study drink supplemented with Xanthohumol + Iso-alpha-Acids (0 mg = Placebo, 0,125 mg + 15 mg , 0,375 mg + 45 mg or 0,75 mg + 90 mg soluble Xanthohumol + Iso-alpha-Acids)
  Arms: Xanthohumol/Iso-alpha-Acids

SUMMARY:
The aim of the present study is to determine the effect of Iso-alpha-Acids and Xanthohumol from hops on the immune response of healthy participants over a timeframe of 6 hours.

DETAILED DESCRIPTION:
In this placebo-controlled crossover study a study drink enriched with either a placebo, Xanthohumol, Iso-alpha Acids or a combination of latter is given to the participants. A washout phase before intervention and between each intervention is introduced. On day one of each intervention blood is drawn in fasted state from each participant. Subsequently the study drink combined with a standardized breakfast is given to the participants followed by blood draws 1, 2, 3, 4 and 6 hours after the consumption of the study drink. To assess the effect of Xanthohumol and Iso-alpha acids or a combination of both, clinical parameters, blood lipids, blood glucose, uric acid and inflammatory markers will be determined. Furthermore, blood cells, isolated from blood samples of each time point, will be stimulated for measuring inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* BMI: >18,5 kg/m² or <30 kg/m²

Exclusion Criteria:

* food intolerances
* food allergies
* chronic inflammatory diseases
* metabolic diseases
* viral or bacterial infections within the last 3 weeks of inclusion
* intake of immunosuppressive medication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in parameters of immune response | 6 hours
  Changes in concentration of interleukin 6 (ng/ml) in cell culture supernatant of stimulated cells.
Changes in parameters of immune response | 6 hours
  Changes in concentration of interleukin 1 beta (ng/ml) in cell culture supernatant of stimulated cells.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No